CLINICAL TRIAL: NCT02251054
Title: Virtual Avatar Coaches for Behavioral Therapy of Patients With Overactive Bladder
Acronym: OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Allen D. Andrade, Staff physician, Miami VA Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WS624459
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Multimedia; Behavioral Therapy
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avatar group (Experimental): Intervention group viewed two avatar coaches: a generic avatar coach (GAC) and a self-avatar, "peer" mentor (SAP).
  Interventions: Other: Avatar group
- No Avatar group (Active Comparator): The control group version (voice only) observed the identical program, including introductions, question asking, narration of animations, delivery of key points, and summary of each section with identical pre-recorded voices without the avatars.
  Interventions: Other: No Avatar group

INTERVENTIONS:
Other: Avatar group — We developed and tested the online program of three multimedia tutorials using the game development and rendering engine (Unity3D, Unity Technologies, San Francisco, CA). This arm saw the tutorials with Avatars.
  Arms: Avatar group
Other: No Avatar group — We developed and tested the online program of three multimedia tutorials using the game development and rendering engine (Unity3D, Unity Technologies, San Francisco, CA). This arm saw the tutorials without Avatars.
  Arms: No Avatar group

SUMMARY:
This study compares the efficacy of embedding avatars into an online self-management program that teaches OAB behavioral therapy on OAB-related quality of life, symptoms, self-efficacy, and adherence versus the same program without avatars

ELIGIBILITY:
Inclusion Criteria:

* age 55 or older
* women living in the community
* who could read and speak English
* urgency (≥3 episodes/24 hrs.) ± urge urinary incontinence
* urinary frequency (≥8 times/24 hrs.)
* nocturia (awakening ≥2 times at night)

Exclusion Criteria:

* hematuria
* abdominal pain
* fever
* cognitive impairment (Mini-Cog < 3)
* positive screen for depression (PHQ2 > 3)
* hearing issues
* uncorrected visual difficulties

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Overactive bladder- health related quality of life (OAB HRQOL) | Baseline and at one, six, and 12 weeks
  The OAB-q is a 33-item measure to assess impact of OAB symptoms on HRQOL. The OAB-q consists of a symptom bother scale and four HRQOL subscales (coping, concern, sleep, and social interaction). All scale scores are transformed to a 0-to-100-point scale, with higher symptom bother scores indicating greater symptom severity, and lower total and subscale scores indicating improvement in HRQOL.27 A 10-point change in these scales indicates a minimal clinically important difference (MCID). The Cronbach alpha coefficient in this study was 0.88.

SECONDARY OUTCOMES:
Perception of Bladder Condition (PPBC) | Baseline and at one, six, and 12 weeks
  The PPBC is a single-item, six-point rating scale of participants subjective assessment of their bladder symptoms, with the question "My bladder causes…" me no (1), very minor (2), minor (3), moderate (4), severe (5), or many severe (6) problems. A two-point negative change indicates an MCID.28
Overactive bladder symptoms | 12 weeks duration
  Participants completed daily bladder diaries data for 12 weeks with information on date, beverage, quantity and time of fluid intake, voiding frequency, voiding volume quantified, urge-related episodes with or without urinary incontinence, and the circumstances of each episode. At each visit, research associates would review bladder diaries to ensure that entries were clear and interpretable. A research associate, blinded to group assignment, scored bladder diaries and managed the data.
Geriatric Self-Efficacy Index for Urinary Incontinence (GSEI) | Baseline and at one, six, and 12 weeks
  The GSEI measures older adults' level of confidence in preventing incontinence episodes. Total scores for the GSEI were computed by summing the scores from each of the 16 items (minimum 0, maximum 10 points per item, range 0-160); a minimum 20-point difference suggests an MCID. The Cronbach alpha coefficient in this study was 0.91.29 We also asked participants at baseline and at one, six, and 12 weeks to describe their confidence in doing pelvic floor muscle exercises: "How confident are you in doing pelvic floor muscle exercises?" and their ability to suppress urge: "How confident are you in suppressing the urge?" on a 100 mm visual analog scales (VAS). The 100 mm VAS was in the range of 0, "not at all confident" to 10, "extremely confident."
Adherence to Pelvic Floor Muscle Exercises (PFMEs) | Baseline and at one, six, and 12 weeks
  Participants were asked how often they had performed PFME in the previous week (0=do not perform, 1=once a week, 2=twice a week once a day, 3=twice a week more than once a day, 4=alternate days once a day, 5= alternate day more than once, 6=every day of the week once a day, 7=every day of the week more than once a day). We also asked about the number of repetitions they did during each exercise session (0=1-2 times, 1=2-4 times, 3=4-6 times, 4=6-8 times, 5=8-10 times, 6=more than 10 times).
Avatar Recognition | At 12 weeks
  The research associate asked participants if they recognized the face of the avatars in the tutorials at 12 weeks with a single question: "Who did the avatar look like?"

CONTACTS AND LOCATIONS:
Overall Officials: Allen D Andrade, MD, Principal Investigator — Miami VAHS
Locations (1):
- Miami VA Healthcare System, Miami, Florida, United States

REFERENCES:
- [Derived] Andrade AD, Anam R, Karanam C, Downey P, Ruiz JG. An overactive bladder online self-management program with embedded avatars: a randomized controlled trial of efficacy. Urology. 2015 Mar;85(3):561-7. doi: 10.1016/j.urology.2014.11.017. Epub 2015 Jan 10. PMID 25586473